CLINICAL TRIAL: NCT03280251
Title: Potentiation of Cognitive Functions in Healthy Elderly by Association of Methylphenidate and Cognitive Training: Proof of Concept Study in Order to Develop a Synergic Symptomatic Treatment for the Cognitive Disorders Before Dementia
Brief Title: Methylphenidate and Cognitive Training in Elderly
Acronym: PACTE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015_81; 2016-005131-32 (EudraCT Number)
Record Dates: First submitted 2017-09-05; First posted 2017-09-12 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers
Keywords: Cognitive disorders; cognitive training; symptomatic treatment; Methylphenidate; elderly
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Methylphenidate and structured cognitive training (Experimental): Methylphenidate (capsules of Ritaline LP 10) encapsulated, 0,3 mg per kg per day during 6 weeks Structured cognitive training with CogniPlus software, twice per week during 6 weeks
  Interventions: Drug: Methylphenidate; Other: CogniPlus software
- Placebo and structured cognitive training (Experimental): Placebo, identical capsules to encapsulated MPH, number of capsules per day identical to MPH during 6 weeks Structured cognitive training with CogniPlus software, twice per week during 6 weeks
  Interventions: Drug: Placebo; Other: CogniPlus software
- Methylphenidate and pseudo cognitive training (Experimental): Methylphenidate (capsules of Ritaline LP 10) encapsulated, 0,3 mg per kg per day during 6 weeks Pseudo cognitive training with 45 minutes documentary videos and 15 minutes quiz, twice per week during 6 weeks
  Interventions: Drug: Methylphenidate; Other: Pseudo cognitive training
- Placebo and pseudo cognitive training (Experimental): Placebo, identical capsules to encapsulated MPH, number of capsules per day identical to MPH during 6 weeks Pseudo cognitive training with 45 minutes documentary videos and 15 minutes quiz, twice per week during 6 weeks
  Interventions: Drug: Placebo; Other: Pseudo cognitive training

INTERVENTIONS:
Drug: Methylphenidate — Methylphenidate (capsules of Ritaline LP 10) encapsulated, 0,3 mg per kg per day during 6 weeks
  Arms: Methylphenidate and pseudo cognitive training; Methylphenidate and structured cognitive training
Drug: Placebo — Placebo, identical capsules to encapsulated MPH, number of capsules per day identical to MPH during 6 weeks
  Arms: Placebo and pseudo cognitive training; Placebo and structured cognitive training
Other: CogniPlus software — Structured cognitive training with CogniPlus software, twice per week during 6 weeks
  Arms: Methylphenidate and structured cognitive training; Placebo and structured cognitive training
Other: Pseudo cognitive training — Pseudo cognitive training with 45 minutes documentary videos and 15 minutes quiz, twice per week during 6 weeks
  Arms: Methylphenidate and pseudo cognitive training; Placebo and pseudo cognitive training

SUMMARY:
Currently, there is no available drug to treat the symptoms of neurodegenerative and vascular cognitive disorders that affect millions of people worldwide.

Methylphenidate is indicated at high dose (1 mg/kg/day) in children having attention deficit and hyperactivity disorder (ADHD) and remains the best cognitive enhancer drug at lower dose. However, there is no proof of efficacy with chronic administration, outside ADHD, and concern remains about long-term cardiac and vascular risks in elderly and particularly in population with vascular risk factors and drug abuse in young people. Moreover, the effect appears to be very limited at the very advanced stage of dementia, for which the neuronal plasticity is too reduced to expect a benefit of training.

Taken all together, we sought to develop a new paradigm of association of both pharmacological and non-pharmacological procedure to enhance the neuronal plasticity in order to expect a persistent effect on slight to mild cognitive disorders with benefit on ecological test (i.e. driving). Finally, short-term treatment would reduce the safety concerns.

The concept will be to prove that low dose of methylphenidate associated with active cognitive training during 6 weeks can improve the cognitive function in healthy aged volunteers with a persistent effect at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Without severe chronic neurological or mental or psychiatric pathology
* Absence of cognitive impairment affecting autonomy (scores on the dementia scale of Mattis> 130 and the IADL = 4)
* Right-handed participant
* Subjects holding driving license B and continuing a driving activity
* Affiliate or beneficiary of a social security scheme
* Subject having signed informed consent
* Subject having agreed to be registered on the National File of Healthy Volunteers
* Patient willing to comply with all procedures of the study and its duration
* No planned changes in lifestyle (nutritional and physical, social interactions) during the life of the protocol

Exclusion Criteria:

* Administrative reasons: impossibility of receiving informed information, inability to participate in the whole study, absence of coverage by the social security system, refusal to sign consent.
* Subject simultaneously participating in another clinical trial or in an exclusion period.
* Subject under tutelage or curatelle.
* Subject during breastfeeding or pregnancy.
* Subject not sufficiently fluent in the French language to understand the instructions necessary to carry out the cognitive tests.
* Subject with uncorrected visual pathology or motor pathology (orthopedic example) likely to interfere with the passing of tests.
* Subject with dependencies pre-existing to medicines, drugs or alcohol.
* Presence of contraindications to MRI: Claustrophobia, Anxiety crisis, Morphotype not allowing access to MRI, metal implant (eg a pacemaker), surgical clips Ferromagnetic, orbital or brain metallic foreign bodies).
* Hypersensitivity to methylphenidate or any other constituents of the product.
* Subject with a personal and / or family history of motor tics and Gilles de la Tourette syndrome.
* Subjects with a previous psychiatric history (based on the semi-structured psychiatric interview with the MINI of DSM IV adapted to DSM V): state, severe depression, severe generalized anxiety, anorexia nervosa or anorexic disorders, suicidal tendencies, psychotic symptoms, severe mood disorders, mania, schizophrenia, psychopathic personality disorder or borderline disorder. Dysthymia and an isolated history of depression do not constitute an exclusion criterion.
* Subjects consuming one or more psychotropic drugs or related products (antidepressants, antipsychotics, antiepileptic drugs, daily use of benzodiazepine anxiolytics or other anxiolytics, vesperal hypnotic intake). A history of taking point hypnotics is not a criterion of exclusion. However, there should be no regular and regular intake in the previous 3 months and less than once a week (ideally, lack of intake would be desirable but would considerably limit the potential for inclusion). They will be asked not to change their habits during the study period.
* Subjects with dysthyroidism or thyrotoxicosis
* Subjects with pre-existing cardiovascular disorders including severe hypertension, heart failure, occlusive arterial disease, angina pectoris, congenital heart disease with hemodynamic repercussions, cardiomyopathy, myocardial infarction, arrhythmias and channelopathies
* Subject with angle-closure glaucoma.
* Significant abnormalities on MRI and EEG according to the investigator's judgment
* Presence of untreated hypertension discovered during screening
* Subject with pheochromocytoma
* Pre-existing cerebrovascular disorders, cerebral aneurysm, vascular abnormalities, including vasculitis or stroke in the subject
* Subjects with hepatic and renal insufficiency
* Obese subject according to WHO classification (BMI> 30)
* Presence of one of the following treatments that cannot be stopped for a period corresponding to 5 half-lives before inclusion: selective and non-selective MAOIs (nialamide and iproniazide, selegiline), other indirect sympathomimetics (phenylpropanolamine, pseudoephedrine, Phenylephrine), halogenated volatile anesthetics, guanethidine and related compounds.
* Treatment with alpha sympathomimetics (oral and / or nasal route) (etilefrin, midodrine, naphazoline, oxymetazoline, tetryzoline, tuaminoheptane, tymazoline), opiates and morphine derivatives. These concomitant treatments are contraindicated at baseline and throughout the study period.
* Subject with leukopathy classified ≥2 on the Fazekas scale

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
The difference of the average response time to a choice task at inclusion and at the end of treatment (after 6 weeks) | 6 weeks after the beginning of the treatment

SECONDARY OUTCOMES:
Change from baseline the composite cognitive functions | Baseline, at 6 weeks, at 12 weeks
  A composite measure of several cognitive functions: attention, executive functions, working memory, verbal and nonverbal episodic memory, visuo-spatial functions
Change from baseline of the results to task on a driving simulator | Baseline, at 6 weeks, at 12 weeks
  A composite measure of task on a driving simulator: travel time, speed parameters(average speed, maintaining the target speed) compliance with the instructions and code of the road (number and type of errors), number of cars doubled, reaction time in analytics.
Behavior Rating Inventory of Executive Function (BRIEF-A) | Baseline, at 6 weeks, at 12 weeks
Hospital Anxiety and Depression scale (HAD) | Baseline, at 6 weeks, at 12 weeks
Number of undesirable effects of treatment | at 2 weeks, at 4 weeks, at 6 weeks, at 12 weeks
Change from baseline the parameters of structured cognitive training (CogniPlus®) | Baseline, at 6 weeks, at 12 weeks
  A composite measure of parameters following : processing speed, inhibition and working memory resources.
Resting state EEG | Baseline, at 6 weeks, at 12 weeks
  EEG with Attentional Network Test and Go / No Go task
resting state functional MRI | Baseline, at 6 weeks, at 12 weeks
  The changes of resting state functional MRI after treatment and cognitive training

CONTACTS AND LOCATIONS:
Overall Officials: David Devos, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France